CLINICAL TRIAL: NCT06582407
Title: Machine Learning Models for Predicting Unforeseen Hospital Admissions or Discharges After Anesthesia
Status: Completed | Type: Observational
Sponsor: HUmani (Network)
Responsible Party: Principal Investigator, Rémi Florquin, Doctor, University of Mons
Other Study IDs: HUmani_ODanesth
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia Complication; Surgery-Complications; Pain, Postoperative
Keywords: anesthesiology; ambulatory surgery; artificial intelligence; machine learning; post operative complication
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ambulatory Patients: Patient undergoing anesthesia in an ambulatory setting.
  Interventions: Other: Mathematical Prediction of unforseen patient reorientation
- Hospitalised Patients: Patient undergoing anesthesia in a hospitalisation setting.
  Interventions: Other: Mathematical Prediction of unforseen patient reorientation

INTERVENTIONS:
Other: Mathematical Prediction of unforseen patient reorientation — The goal of this project is to develop models to predict in the preoperative period which patients will require hospital admission after ambulatory surgery or unforeseen hospital discharge after surgery

SUMMARY:
Unexpected hospital admissions after ambulatory surgery not only bring discomfort to patients but also causes a decrease in the efficiency of the healthcare system. In addition, unanticipated patient's orientation carry the risk of unsuitable post operative orders. The hypothesis of this project is that artificial intelligence models will outperform traditional models in predicting which patients will require hospital admission after ambulatory surgery or unforeseen hospital discharge after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing anesthesia for a therapeutic or diagnostic procedure

Exclusion Criteria:

* Incomplete informatic data
* Error in the encoding system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospitalized or outpatient patients who have undergone anesthesia for a diagnostic or therapeutic procedure, in a scheduled or emergency condition, in the institution's hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 68683 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of patient reorientation | On the day of the operation
  Rate of unforeseen hospital admission after an ambulatory surgery and rate of discharge after an hospitalised surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Florquin, MD, Principal Investigator — Université de Mons, Belgium
Locations (1):
- Université de Mons, Mons, Belgium

IPD SHARING:
Plan to Share IPD: No
The investigators are not authorized to publish sensitive data by decision of the ethics committee